CLINICAL TRIAL: NCT02283827
Title: Phase I, Open-label Drug Interaction Study Between Eslicarbazepine Acetate 1200mg and Phenytoin 300 mg Following Multiple Dose Administrations in Healthy Male Volunteers
Brief Title: Open-label Drug Interaction Study Between Eslicarbazepine Acetate and Phenytoin.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-121
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A BIA 2-093 + Phenytoin (PHT) (Experimental): Day 1 to 2: Pre-treatment 1: 600 mg ESL Day 3 to 8: Treatment 1: 1200 mg ESL Day 9 to 10: Treatment 1 + Pre-treatment 2: 1200 mg ESL+ 100 mg PHT Day 11 to 27: Treatment 1 + Treatment 2: 1200 mg ESL + 300 mg PHT
  Interventions: Drug: BIA 2-093; Drug: Phenytoin
- Group B BIA 2-093 + Phenytoin (PHT) (Experimental): Day 1 to 2: Pre-treatment 2: 100 mg PHT Day 3 to 8: Treatment 2: 300 mg PHT Day 9 to 10: Treatment 2 + Pre-treatment 1: 300 mg PHT + 600 mg ESL Day 11 to 27: Treatment 1 + Treatment 2: 1200 mg ESL + 300 mg PHT
  Interventions: Drug: BIA 2-093; Drug: Phenytoin

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: Eslicarbazepine acetate; ESL
Drug: Phenytoin
  Other Names: PHT

SUMMARY:
Single centre, open-label, multiple doses, two parallel study groups each receiving two formulations in a one-sequence design

DETAILED DESCRIPTION:
Single centre, open-label, multiple doses, two parallel study groups each receiving two formulations in a one-sequence design:

Group A: Pre-treatment with ESL, treatment with ESL and ascending doses of phenytoin (PHT) in last phases;

Group B: Pre-treatment with PHT, treatment with PHT and ascending doses of ESL in last phases

ELIGIBILITY:
Inclusion Criteria:

* Availability of volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
* Non-black male aged of at least 18 years but not older than 45 years with a body mass index (BMI) greater than or equal to 19 and below 30 kg/m2
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance (laboratory tests are presented in section 6.1.1.3)
* Healthy according to the medical history, laboratory results and physical examination
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day, and an ex-smoker is defined as someone who completely stopped smoking for at least 12 months before day 1 of this study

Exclusion Criteria:

* Significant history of hypersensitivity to phenytoin, eslicarbazepine, oxcarbazepine, carbamazepine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability, including but not limited to cholecystectomy
* Presence of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of significant heart disease or disorder according to ECG
* Presence or history of significant central nervous system disorder like convulsion or depression
* Hemoglobin count below 135 g/L (at screening)
* Use of valproic acid in the previous 7 days prior to Day 1 of the study.
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids,phenytoin and rifampin), in the previous 28 days before Day 1 of this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A BIA 2-093 + Phenytoin (PHT): Day 1 to 2: Pre-treatment 1: ESL 600 mg Day 3 to 8: Treatment 1:1200 mg ESL Day 9 to 10: Treatment 1 + Pre-treatment 2: 1200 mg ESL+ PHT 100 mg Day 11 to 27: Treatment 1 + Treatment 2: 1200 mg ESL + PHT 300 mg
- Group B BIA 2-093 + Phenytoin (PHT): Day 1 to 2: Pre-treatment 2: PHT 100 mg Day 3 to 8: Treatment 2: PHT 300 mg Day 9 to 10: Treatment 2 + Pre-treatment 1: PHT 300 mg
  + ESL 600 mg Day 11 to 27: Treatment 1 + Treatment 2: 1200 mg ESL + PHT 300 mg
Period: Overall Study
Arm/Group | Group A BIA 2-093 + Phenytoin (PHT) | Group B BIA 2-093 + Phenytoin (PHT)
Started | 16 | 16
Completed | 15 | 13
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group A BIA 2-093 + Phenytoin (PHT): Pre-treatment: 600 mg ESL, 2 days; Treatment 1: 1200 mg ESL 6 days Treatment 2: 1200 mg ESL and PHT 100 mg for 2 days Treatment 3: 1200 mg ESL and PHT 300 mg for17 days
- Group B BIA 2-093 + Phenytoin (PHT): Pre-treatment: 100 mg PHT for 2 days; Treatment 1: 300 mg PHT 6 days; Treatment 2: 600 mg ESL + PHT 300 mg for 2 days; Treatment 3: 1200 mg ESL and PHT 300 mg for 17 days
- Total: Total of all reporting groups
Arm/Group | Group A BIA 2-093 + Phenytoin (PHT) | Group B BIA 2-093 + Phenytoin (PHT) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax - the Maximum Plasma Concentration
Description: BIA 2-194 and BIA 2-195 are metabolites of eslicarbazepine acetate
Time Frame: Day 8 and 27: within 5 minutes prior to dosing and 0.5,1,1.5,2,2.5,3,3.5,4,6,9,12,16 and 24 hours after drug administration
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 2-093 + Phenytoin: Phenytoin - PHT; BIA 2-093 - ESL, Eslicarbazepine
- BIA 2-093: BIA 2-093 - ESL, Eslicarbazepine
Arm/Group | BIA 2-093 + Phenytoin | BIA 2-093
Number analyzed (Participants) | 28 | 15
ng/mL
  Cmax (BIA 2-194) | 16350.6 (2060.2) | 23806.5 (3047.2)
  Cmax (BIA 2-195) | 976.9 (194.4) | 954.3 (189.9)
  Cmax (PHT) | 12868.5 (6292.7) | 9405.1 (3621)

2. Secondary Outcome: AUC0-t - the Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time
Description: AUC0-t - the Area Under the Plasma Concentration-time Curve From Time Zero to the Last Sampling Time
  BIA 2-194 and BIA 2-195 are metabolites of eslicarbazepine acetate
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- BIA 2-093 + Phenytoin (PHT): Phenytoin - PHT BIA 2-093 - ESL, Eslicarbazepine
Arm/Group | BIA 2-093 + Phenytoin (PHT) | BIA 2-093
Number analyzed (Participants) | 28 | 15
ng*h/mL
  AUC0-t (BIA 2-194) | 251055.2 (34143.1) | 371574.9 (43474.3)
  AUC0-t (BIA 2-195) | 19471.2 (4069.5) | 20675.0 (4362.4)
  AUC0-t (PHT) | 264784.8 (137688.1) | 186826.5 (81643.2)

3. Secondary Outcome: Tmax - the Time of Occurrence of Cmax
Description: BIA 2-194 and BIA 2-195 are metabolites of eslicarbazepine acetate
Time Frame: as for outcome 1
Measure: Median (Standard Deviation); unit: hours
Arm/Group | BIA 2-093 + Phenytoin (PHT) | BIA 2-093
Number analyzed (Participants) | 28 | 15
hours
  Tmax (BIA 2-194) | 3.00 (1.02) | 2.50 (0.95)
  Tmax (BIA 2-195) | 9.00 (1.49) | 9.00 (4.03)
  Tmax (PHT) | 4.00 (1.96) | 4.00 (2.35)

ADVERSE EVENTS:
Time Frame: Day 8 was used for BIA 2-093 group and Day 27 was used for BIA 2-093 + Phenytoin group
Groups:
- BIA 2-093 600 mg; BIA 2-093 1200 mg: BIA 2-093 - ESL, Eslicarbazepine
- BIA 2-093 1200 mg + Phenytoin 100 mg; BIA 2-093 1200 mg + Phenytoin 300 mg; BIA 2-093 600 mg + Phenytoin 300 mg: Phenytoin - PHT BIA 2-093 - ESL, Eslicarbazepine
- Phenytoin 100 mg: Phenytoin - PHT 100 mg
- Phenytoin 300 mg: Phenytoin - PHT 300 mg
Arm/Group | BIA 2-093 600 mg | BIA 2-093 1200 mg | BIA 2-093 1200 mg + Phenytoin 100 mg | BIA 2-093 1200 mg + Phenytoin 300 mg | Phenytoin 100 mg | Phenytoin 300 mg | BIA 2-093 600 mg + Phenytoin 300 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/32 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 3/16 | 12/16 | 7/16 | 27/32 | 7/16 | 10/16 | 8/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 2-093 600 mg (N=16) | BIA 2-093 1200 mg (N=16) | BIA 2-093 1200 mg + Phenytoin 100 mg (N=16) | BIA 2-093 1200 mg + Phenytoin 300 mg (N=32) | Phenytoin 100 mg (N=16) | Phenytoin 300 mg (N=16) | BIA 2-093 600 mg + Phenytoin 300 mg (N=16)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrheoa (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 3 | 1 | 3 | 0 | 1 | 1
Feeling drunk (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hot flush (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 10 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 3 | 2 | 8 | 1 | 1 | 0
Insomnia (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Nervous system disorders) | 1 | 3 | 0 | 4 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 7 | 4 | 11 | 6 | 1 | 3
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Erection increased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry throat (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysguesia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tooth abscess (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
white blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other